CLINICAL TRIAL: NCT00630331
Title: A Phase III, Randomized, Observer-Blind, Placebo-Controlled, Multicenter Study to Assess Clinical Efficacy of a Cell-Derived Subunit Influenza Vaccine and an Egg-Derived Subunit Influenza Vaccine in the 2007-2008 Influenza Season in Healthy Adult Subjects
Brief Title: Efficacy Study of Two Influenza Vaccines and Placebo in Healthy Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V58P13; 2007-002871-15; 11580
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Influenza
Keywords: Influenza; Flu; Cell Culture-Derived; Egg-Derived; Healthy Adults; Efficacy; Safety; Immunogenicity; Trivalent; Inactivated; Influenza-Like Illness; Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- CCI (Experimental): Subjects received one dose of cell culture-derived influenza vaccine.
  Interventions: Biological: Cell culture-derived influenza vaccine
- IVV (Experimental): Subjects received one dose of the trivalent egg-derived influenza vaccine.
  Interventions: Biological: Egg-derived influenza virus vaccine
- Placebo (Placebo Comparator): Subjects received one dose of phosphate buffered solution (PBS).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Cell culture-derived influenza vaccine — One dose (0.5 mL) of cell culture-derived influenza vaccine, administered in the deltoid muscle.
  Arms: CCI
Biological: Egg-derived influenza virus vaccine — One dose (0.5 mL) of the trivalent egg-derived influenza virus vaccine, administered in the deltoid muscle.
  Arms: IVV
Biological: Placebo — One dose (0.5 mL) of phosphate buffered solution.
  Arms: Placebo

SUMMARY:
The present study will evaluate clinical efficacy, safety, tolerability and immunogenicity of both Novartis Vaccines' cell-derived influenza vaccine and egg-derived influenza vaccine in healthy adults 18 to 49 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. subjects 18 to 49 years of age;
2. in good health as determined by medical history and physical examination;
3. able and willing to provide written informed consent prior to any study procedure;
4. able to comply with all study procedures, including availability and willingness to be actively followed throughout the ensuing influenza season with weekly telephone calls and to comply with the need for prompt collection of nasal and throat specimens in the event of influenza symptoms.

Exclusion Criteria:

1. history of anaphylaxis or serious reaction after administration of any vaccine, or hypersensitivity to eggs, egg protein, chicken feathers, influenza viral protein, neomycin, kanamycin, or any other vaccine component, chemically related substance, or component of the potential packaging materials;
2. any health condition for which the inactivated vaccine is recommended by the Advisory Committee on Immunization Practices (ACIP) including chronic diseases of the pulmonary or cardiovascular systems (including asthma), chronic metabolic diseases (including diabetes), renal dysfunction, hemoglobinopathies, immune deficiency disease (including HIV infection) or on-going immunosuppressive therapy;
3. employment in professions prone to influenza transmission to or from high-risk populations (this exclusion specifically includes nurses, physicians, all other healthcare workers with direct patient contact; and police, fire, and rescue personnel); or living in the same household as an immunocompromised person;
4. history of Guillain-Barré syndrome;
5. bleeding diathesis;
6. receipt of another investigational agent within 90 days prior to enrollment in the study or before completion of the safety follow-up period in another study, whichever is longer, and unwilling to refuse participation in another clinical study through the end of the study;
7. receipt of another vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to Visit 1;
8. laboratory-confirmed influenza disease within 6 months prior to Visit 1;
9. receipt of an influenza vaccine within 6 months prior to Visit 1 or plans to receive influenza vaccine outside of this study;
10. experienced a temperature (≥100.0°F / ≥37.8°C) and/or any acute illness within 3 days prior to study vaccination;
11. pregnant or breast-feeding female;
12. if female of childbearing potential and sexually active, has not used any of the birth control methods detailed in the section entitled "Females of Childbearing Potential" for at least 2 months prior to study entry;
13. if female of childbearing potential and sexually active, refusal to use a reliable contraceptive method as detailed in the section entitled "Females of Childbearing Potential" during the first 3 weeks after vaccination;
14. research staff directly involved with the clinical study or family members or household members of research staff. Research staff are individuals with direct or indirect contact with study subjects, or study site personnel who have access to any study documents containing subject information. This would include receptionists, persons scheduling appointments or making screening calls, regulatory specialists, laboratory technicians, etc.;
15. any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives or with the safety of the study subject.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11404 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (56):
- United States (17):
  - Site 14, Denver, Colorado
  - Site 15, Pembroke Pines, Florida
  - Site 17, South Miami, Florida
  - Site 13, Lenexa, Kansas
  - Site 2, Bardstown, Kentucky
  - Site 1, St Louis, Missouri
  - Site 4, Edison, New Jersey
  - Site 10, Binghamton, New York
  - Site 5, Endwell, New York
  - Site 16, Winston-Salem, North Carolina
  - Site 11, Warwick, Rhode Island
  - Site 12, Anderson, South Carolina
  - Site 9, Austin, Texas
  - Site 8, Dallas, Texas
  - Site 7, Salt Lake City, Utah
  - Site 3, Salt Lake City, Utah
  - Site 6, Burke, Virginia
- Finland (15):
  - Site 25, Espoo
  - Site 26, Helsinki
  - Site 27, Helsinki
  - Site 33, Jarvenpaa
  - Site 35, Kokkola
  - Site 34, Kotka
  - Site 30, Kuopio
  - Site 22, Lahti
  - Site 31, Oulu
  - Site 23, Pori
  - Site 32, Seinäjoki
  - Site 21, Tampere
  - Site 24, Turku
  - Site 28, Vantaa
  - Site 29, Vantaa
- Poland (24):
  - Site 49, Bydgoszcz
  - Site 62, Gmina Końskie
  - Site 53, Gniewkowo
  - Site 59, Katowice
  - Site 63, Kielce
  - Site 57, Krakow
  - Site 41, Krakow
  - Site 43, Krakow
  - Site 42, Krakow
  - Site 50, Krakow
  - Site 44, Lubartów
  - Site 45, Lublin
  - Site 65, Oleśnica
  - Site 47, Olsztyn
  - Site 48, Olsztyn
  - Site 46, Olsztyn
  - Site 58, Radziszów
  - Site 61, Ruda Śląska
  - Site 60, Rzeszów
  - Site 52, Warsaw
  - Site 54, Wąbrzeźno
  - Site 55, Wilkowice
  - Site 64, Wroclaw
  - Site 51, Łodź

REFERENCES:
- [Result] Frey S, Vesikari T, Szymczakiewicz-Multanowska A, Lattanzi M, Izu A, Groth N, Holmes S. Clinical efficacy of cell culture-derived and egg-derived inactivated subunit influenza vaccines in healthy adults. Clin Infect Dis. 2010 Nov 1;51(9):997-1004. doi: 10.1086/656578. PMID 20868284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at multiple centres in the US, Poland and Finland.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- CCI Vaccine: One dose of cell culture-derived influenza vaccine.
- IVV Vaccine: One dose of the trivalent egg-derived influenza virus vaccine.
- Placebo: One dose of phosphate buffered solution (PBS).
Period: Overall Study
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Started | 3828 | 3676 | 3900
Completed | 3622 | 3510 | 3712
Not Completed | 206 | 166 | 188
Not completed — Death | 2 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 7 | 5
Not completed — Lost to Follow-up | 175 | 143 | 170
Not completed — Inappropriate enrollment | 3 | 6 | 3
Not completed — Unable to classify | 9 | 4 | 3
Not completed — Protocol Violation | 4 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo | Total
Number analyzed (Participants) | 3828 | 3676 | 3900 | 11404
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (10.1) | 33.0 (10.2) | 32.7 (10.2) | 32.8 (10.2)
Sex/Gender, Customized [Number; unit: Subjects] — Baseline Characteristics are reported for the Enrolled Population. For 3 of 11404 subjects, data on gender was not reported. Therefore, these data are not available.
  Subjects
    Female | 2088 | 2026 | 2176 | 6290
    Male | 1740 | 1649 | 1722 | 5111
    Not Available | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Culture-Confirmed Influenza Illness Caused by Vaccine-like Strains
Description: The vaccine efficacy of CCI and IVV vaccines was estimated relative to Placebo group as the number of subjects prevented against virus-confirmed symptomatic influenza illness caused by each of three vaccine-like virus strains.
Time Frame: 6 Months
Population: Analysis was performed on per protocol (PP) efficacy population i.e. the subjects in the exposed efficacy population who correctly received the vaccine and provided evaluable swab samples at the relevant time points.
Measure: Number; unit: Subjects
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 3776 | 3638 | 3843
Subjects
  Overall | 7 | 9 | 44
  A/Wisconsin/67/2005 (H3N2)-like | 2 | 1 | 0
  A/Solomon Islands/3/2006 (H1N1)-like | 5 | 8 | 43
  B/Malaysia/2506/2004-like | 0 | 0 | 1
Statistical Analysis 1: Comparison: CCI Vaccine vs Placebo; Vaccine efficacy (VE) of CCI vaccine vs. Placebo (Overall) Simultaneous one-sided 97.5% confidence interval (CI) for the VE of CCI vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p < 0.001, Sidak-corrected score CI — Adjusted p-values are from score statistic with Sidak correction testing the null hypothesis that the VE of CCI vs. placebo is <= 40% (the relative risk, >= 0.60). If adjusted p-value is <0.025, then the comparison is statistically significant; Vaccine Efficacy = 83.8, 97.5% CI 1-sided [lower limit 61.0]
Statistical Analysis 2: Comparison: CCI Vaccine vs Placebo; Vaccine efficacy (VE) of CCI vaccine vs. Placebo for A/H1N1 strain Simultaneous one-sided 97.5% confidence interval (CI) for the VE of CCI vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p < 0.001, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 88.2, 97.5% CI 1-sided [lower limit 67.4]
Statistical Analysis 3: Comparison: CCI Vaccine vs Placebo; Vaccine efficacy (VE) of CCI vaccine vs. Placebo for A/H3N2 strain. Simultaneous one-sided 97.5% confidence interval (CI) for the VE of CCI vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p = 0.999, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; For strain A/H3N2, the vaccine efficacy of the CCI vaccine vs. placebo was not evaluable since no influenza case was observed in the placebo group
Statistical Analysis 4: Comparison: CCI Vaccine vs Placebo; Vaccine efficacy (VE) of CCI vaccine vs. Placebo for B strain Simultaneous one-sided 97.5% confidence interval (CI) for the VE of CCI vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p = 0.394, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 100, 97.5% CI 1-sided [lower limit -410]
Statistical Analysis 5: Comparison: IVV Vaccine vs Placebo; Vaccine efficacy (VE) of IVV vaccine vs. Placebo (Overall) Simultaneous one-sided 97.5% confidence interval (CI) for the VE of IVV vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p = 0.004, Sidak-corrected score CI — Adjusted p-values are from score statistic with Sidak correction testing the null hypothesis that the VE of IVV vs. placebo is <= 40% (the relative risk, >= 0.60). If adjusted p-value is <0.025, then the comparison is statistically significant; Vaccine Efficacy = 78.4, 97.5% CI 1-sided [lower limit 52.1]
Statistical Analysis 6: Comparison: IVV Vaccine vs Placebo; Vaccine efficacy (VE) of IVV vaccine vs. Placebo for A/H1N1 strain Simultaneous one-sided 97.5% confidence interval (CI) for the VE of IVV vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p = 0.002, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 80.3, 97.5% CI 1-sided [lower limit 54.7]
Statistical Analysis 7: Comparison: IVV Vaccine vs Placebo; Vaccine efficacy (VE) of IVV vaccine vs. Placebo for A/H3N2 strain. Simultaneous one-sided 97.5% confidence interval (CI) for the VE of IVV vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p = 0.992, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; For strain A/H3N2, the vaccine efficacy of the IVV vaccine vs. placebo was not evaluable since no influenza case was observed in the placebo group
Statistical Analysis 8: Comparison: IVV Vaccine vs Placebo; Vaccine efficacy (VE) of IVV vaccine vs. Placebo for B strain Simultaneous one-sided 97.5% confidence interval (CI) for the VE of IVV vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p = 0.400, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 100, 97.5% CI 1-sided [lower limit -429.4]

2. Secondary Outcome: Number of Subjects With Culture-confirmed Influenza Illness Caused by Non-Vaccine Like Strains
Description: The vaccine efficacy of CCI and IVV vaccines was estimated relative to placebo group as the number of subjects prevented against virus-confirmed symptomatic influenza A or B illness caused by non-vaccine-like strains.
Time Frame: 6 Months
Population: Analysis was done on PP efficacy population.
Measure: Number; unit: Subjects
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 3776 | 3638 | 3843
Subjects
  Overall | 30 | 29 | 74
  A/H3N2 | 0 | 2 | 8
  A/H1N1 | 1 | 0 | 8
  B | 29 | 27 | 59
Statistical Analysis 1: Comparison: CCI Vaccine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.078, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 58.7, 97.5% CI 1-sided [lower limit 33.5]
Statistical Analysis 2: Comparison: CCI Vaccine vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.104, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 87.3, 97.5% CI 1-sided [lower limit 4.6]
Statistical Analysis 3: Comparison: CCI Vaccine vs Placebo; Vaccine efficacy (VE) of CCI vaccine vs. Placebo for A/H3N2 strain Simultaneous one-sided 97.5% confidence interval (CI) for the VE of CCI vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p = 0.030, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 100, 97.5% CI 1-sided [lower limit 36.3]
Statistical Analysis 4: Comparison: CCI Vaccine vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.376, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 50.0, 97.5% CI 1-sided [lower limit 17.5]
Statistical Analysis 5: Comparison: IVV Vaccine vs Placebo; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.085, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 58.6, 97.5% CI 1-sided [lower limit 32.9]
Statistical Analysis 6: Comparison: IVV Vaccine vs Placebo; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; p = 0.033, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 100, 97.5% CI 1-sided [lower limit 33.9]
Statistical Analysis 7: Comparison: IVV Vaccine vs Placebo; Vaccine efficacy (VE) of IVV vaccine vs. Placebo for A/H3N2 strain Simultaneous one-sided 97.5% confidence interval (CI) for the VE of IVV vaccine relative to Placebo was based on the Sidak-corrected score CIs for the two relative risks; Test type: Superiority or Other; p = 0.265, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 73.6, 97.5% CI 1-sided [lower limit -30.0]
Statistical Analysis 8: Comparison: IVV Vaccine vs Placebo; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.319, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 51.7, 97.5% CI 1-sided [lower limit 19.4]

3. Secondary Outcome: Number of Subjects With Influenza Caused by Vaccine-like and Non-vaccine-like Strains
Description: The vaccine efficacy of CCI and IVV vaccines was estimated relative to placebo as the number of subjected prevented against virus-confirmed symptomatic influenza A or B illness caused by vaccine-like and non-vaccine-like strains.
Time Frame: 6 Months
Population: Analysis was done on PP efficacy population.
Measure: Number; unit: Subjects
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 3776 | 3638 | 3843
Subjects
  Overall | 42 | 49 | 140
  A/H3N2 | 6 | 12 | 25
  A/H1N1 | 6 | 10 | 57
  B | 30 | 27 | 61
Statistical Analysis 1: Comparison: CCI Vaccine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 69.5, 97.5% CI 1-sided [lower limit 55.0]
Statistical Analysis 2: Comparison: CCI Vaccine vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 89.3, 97.5% CI 1-sided [lower limit 73.0]
Statistical Analysis 3: Comparison: CCI Vaccine vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.040, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 75.6, 97.5% CI 1-sided [lower limit 35.1]
Statistical Analysis 4: Comparison: CCI Vaccine vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.37, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 1]; Vaccine Efficacy = 49.9, 97.5% CI 1-sided [lower limit 18.2]
Statistical Analysis 5: Comparison: IVV Vaccine vs Placebo; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.003, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 63.0, 97.5% CI 1-sided [lower limit 46.7]
Statistical Analysis 6: Comparison: IVV Vaccine vs Placebo; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; p < 0.001, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 81.5, 97.5% CI 1-sided [lower limit 60.9]
Statistical Analysis 7: Comparison: IVV Vaccine vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.53, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 49.3, 97.5% CI 1-sided [lower limit -9.0]
Statistical Analysis 8: Comparison: IVV Vaccine vs Placebo; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.26, Sidak-corrected score CI — [p-value comment as in outcome 1, analysis 5]; Vaccine Efficacy = 53.2, 97.5% CI 1-sided [lower limit 22.2]

4. Secondary Outcome: Influenza-Associated Days in Bed, All Subjects
Description: The number of subjects in this analysis included all subjects in the per protocol efficacy population.
Time Frame: 6 Months
Population: Analysis was done on the PP efficacy population.
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 3775 | 3638 | 3837
Number of Days | 0.04 (0.496) | 0.04 (0.404) | 0.12 (0.777)

5. Secondary Outcome: Influenza-Associated Days in Bed, Subset of Subjects With Virus-Confirmed- Influenza
Description: The analysis was done among the subset of subjects in the per protocol efficacy population who had culture-confirmed influenza.
Time Frame: 6 Months
Population: Analysis was done on PP efficacy population.
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 180 | 230 | 332
Number of Days | 3.9 (2.62) | 2.9 (1.98) | 3.4 (2.4)

6. Secondary Outcome: Number Of Medical Visits (Inpatient and Outpatient) Due to Influenza Illness or Symptoms of Influenza, All Subjects
Description: The number of subjects in this analysis included all subjects in the per protocol efficacy population.
Time Frame: 6 Months
Population: Analysis was done of PP efficacy population.
Measure: Mean (Standard Deviation); unit: Number of Medical Visits
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 3775 | 3638 | 3838
Number of Medical Visits | 0.01 (0.138) | 0.01 (0.134) | 0.03 (0.262)

7. Secondary Outcome: Number of Medical Visits (Inpatient and Outpatient), Subset of Subjects With Virus-Confirmed-Influenza
Description: as for outcome 5
Time Frame: 6 Months
Population: Analysis was done of PP efficacy population.
Measure: Mean (Standard Deviation); unit: Number of Medical Visits
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 180 | 230 | 332
Number of Medical Visits | 0.8 (0.92) | 0.6 (1.0) | 0.8 (1.16)

8. Secondary Outcome: Number of Days of Usual Activity (i.e. Job, School,Household/Family/Community Activities) Lost Due to Influenza Disease, All Subjects
Description: The number of subjects in this analysis included all subjects in the per protocol efficacy population.
Time Frame: 6 Months
Population: Analysis was done on PP efficacy population.
Measure: Mean (Standard Deviation); unit: Numebr of Days of Usual Activity Lost
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 3775 | 3638 | 3837
Numebr of Days of Usual Activity Lost | 0.06 (0.635) | 0.05 (0.605) | 0.16 (1.006)

9. Secondary Outcome: Number of Days of Usual Activity (i.e. Job, School,Household/Family/Community Activities) Lost, Subset of Subjects With Virus-Confirmed-Influenza
Description: as for outcome 5
Time Frame: 6 Months
Population: Analysis was done on PP efficacy population.
Measure: Mean (Standard Deviation); unit: Numebr of Days of Usual Activity Lost
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 180 | 230 | 332
Numebr of Days of Usual Activity Lost | 5.1 (3.41) | 4.0 (3.4) | 4.6 (3.45)

10. Secondary Outcome: Percentages of Subjects Who Achieved HI Titers ≥40 After One Vaccination of Either Cell-culture Derived or Egg-derived Influenza Vaccine or Placebo
Description: Immunogenicity was measured as the percentage of subjects achieving HI titers ≥40 at baseline (day 1) and three weeks after (day 22) one vaccination of either cell-culture or egg-derived vaccine or placebo for each of the three influenza vaccine strains (A/H1N1, A/H3N2 and B), evaluated using hemagglutination inhibition (HI) egg-derived antigen assay. This criterion is met according to US (CBER) guideline if the lower limit of the two-sided 95% CI for the percentage of subjects achieving HI titers ≥40 is ≥70%.
Time Frame: Before vaccination (day 1) and three weeks after vaccination (day 22)
Population: Analysis was done on a subset of subjects who constituted the PP immunogenicity population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 228 | 695 | 55
Percentages of subjects
  A/H1N1 - Day 1 | 48 [42 to 55] | 53 [49 to 57] | 60 [46 to 73]
  A/H1N1 - Day 22 | 99 [97 to 100] | 98 [97 to 99] | 60 [46 to 73]
  A/H3N2 - Day 1 | 63 [57 to 69] | 58 [54 to 61] | 71 [57 to 82]
  A/H3N2 - Day 22 | 99 [97 to 100] | 99 [98 to 100] | 65 [51 to 78]
  B - Day 1 | 25 [20 to 31] | 23 [20 to 27] | 22 [12 to 35]
  B - Day 22 | 78 [72 to 83] | 92 [90 to 94] | 22 [12 to 35]

11. Secondary Outcome: Percentages of Subjects Achieving Seroconversion After One Vaccination of Either Cell-culture Derived or Egg-derived Influenza Vaccine or Placebo
Description: As per the CBER guideline, seroconversion is defined as the percentage of subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or in subjects with prevaccination HI titer ≥10, a ≥4-fold increase in postvaccination HI antibody titer. According to CBER criteria, the lower limit of the two-sided 95% CI for the percentage of subjects achieving seroconversion for HI antibody titer at day 22 met exceeded 40%.
Time Frame: Three weeks after vaccination (day 22)
Population: Analysis was done on a subset of subjects who constituted the PP immunogenicity population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 228 | 695 | 55
Percentages of subjects
  A/H1N1 | 78 [72 to 83] | 75 [71 to 78] | 0 [0 to 6]
  A/H3N2 | 59 [53 to 66] | 68 [64 to 71] | 0 [0 to 6]
  B | 51 [45 to 58] | 68 [65 to 72] | 0 [0 to 6]

12. Secondary Outcome: Number of Subjects Reported Solicited Local and Systemic Reactions up to 7 Days After Vaccination
Description: The solicited local and systemic reactogenicity were collected up to 7 days after vaccination for all three vaccine groups.
Time Frame: Up to 7 days post vaccination
Population: Analysis was done on Safety population i.e. all subjects in the exposed population who provide post vaccination safety data.
Measure: Number; unit: Subjects
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Number analyzed (Participants) | 3813 | 3669 | 3894
Subjects
  Injection site Pain: number analyzed (Participants) | 3813 | 3668 | 3894
  Injection site Pain | 1158 | 893 | 375
  Injection site Erythema: number analyzed (Participants) | 3813 | 3668 | 3894
  Injection site Erythema | 510 | 492 | 391
  Injection site Induration: number analyzed (Participants) | 3813 | 3668 | 3894
  Injection site Induration | 239 | 207 | 101
  Injection site Ecchymosis: number analyzed (Participants) | 3813 | 3668 | 3894
  Injection site Ecchymosis | 143 | 110 | 147
  Injection site Swelling: number analyzed (Participants) | 3813 | 3667 | 3894
  Injection site Swelling | 218 | 181 | 103
  Chills | 210 | 211 | 223
  Malaise: number analyzed (Participants) | 3813 | 3669 | 3893
  Malaise | 290 | 259 | 237
  Myalgia: number analyzed (Participants) | 3813 | 3669 | 3893
  Myalgia | 450 | 364 | 275
  Arthralgia: number analyzed (Participants) | 3813 | 3669 | 3893
  Arthralgia | 108 | 111 | 125
  Headache: number analyzed (Participants) | 3813 | 3669 | 3893
  Headache | 564 | 551 | 592
  Sweating: number analyzed (Participants) | 3812 | 3669 | 3893
  Sweating | 124 | 122 | 120
  Fatigue: number analyzed (Participants) | 3812 | 3669 | 3893
  Fatigue | 390 | 404 | 384
  Fever (>= 38 C) | 27 | 21 | 15
  Oral Temp. (< 38 C) | 3786 | 3648 | 3879
  Stayed home due to Reactions (N=3781, 3651, 3867): number analyzed (Participants) | 3781 | 3651 | 3867
  Stayed home due to Reactions (N=3781, 3651, 3867) | 42 | 62 | 42
  Analgesic medicines used: number analyzed (Participants) | 3810 | 3665 | 3892
  Analgesic medicines used | 394 | 397 | 386

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were collected throughout the study period (i.e., 6 months).
Description: The analysis was done on the safety population.
Arm/Group | CCI Vaccine | IVV Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 42/3813 | 35/3669 | 38/3894
Other Adverse Events (participants affected / at risk) | 1949/3813 | 1703/3669 | 1387/3894
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CCI Vaccine (N=3813) | IVV Vaccine (N=3669) | Placebo (N=3894)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal Obstructon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peritoneal Cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary Duct Inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary Gland Calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting in Pregnancy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholangitis Sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Breast Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Perirectal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Chest Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Adenocarcinoma of the Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carcinoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tethered Cord Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
Delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
Acute Stress Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Borderline Personality Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder Prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Polycystic Ovaries (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Homicide (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Aortic Valve Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Appendicetomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Knee Operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Medical Device Removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Nasal Septal Operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Rhinoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tendon Operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Varicose Vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CCI Vaccine (N=3813) | IVV Vaccine (N=3669) | Placebo (N=3894)
Chills (General disorders) | 212 | 212 | 225
Fatigue (General disorders) | 390 | 404 | 386
Injection Site Erythema (General disorders) | 510 | 492 | 391
Injection Site Induration (General disorders) | 239 | 207 | 101
Injection Site Pain (General disorders) | 1158 | 893 | 375
Injection Site Swelling (General disorders) | 218 | 181 | 103
Malaise (General disorders) | 290 | 260 | 238
Myalgia (Musculoskeletal and connective tissue disorders) | 451 | 369 | 278
Headache (Nervous system disorders) | 571 | 554 | 597

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No